CLINICAL TRIAL: NCT00874406
Title: Preoperative Transhepatic Arterial Chemotherapy in the Treatment of Liver Metastasis of Resectable Colorectal Cancer
Brief Title: Preoperative Transhepatic Arterial Chemotherapy (TAC) in the Treatment of Liver Metastasis of Resectable Colorectal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Xujianmin, Zhongshan hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-04
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2009-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; liver metastasis; neoadjuvant chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Triamcinolone; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): transhepatic arterial chemotherapy (TAC) were given 7 days before liver metastasis resection. Adjuvant folfox4 chemotherapy was done within 28 days after surgery.
  Interventions: Drug: tac + folfox4
- 2 (Active Comparator): Liver metastasis resection was done without TAC. Adjuvant folfox4 chemotherapy was done within 28 days after surgery.
  Interventions: Drug: folfox4

INTERVENTIONS:
Drug: tac + folfox4 — tac: oxaliplatin 100mg + fudr 1g + mmc 10mg 7 days later： operation within 28 days after operation: folfox4
  Arms: 1
Drug: folfox4 — folfox4 will be done within 28 days after liver resection
  Arms: 2

SUMMARY:
The purpose of this study is to investigate whether preoperative TAC is able to improve progression free survival and overall survival in patients receiving liver metastasis resection of colorectal cancer.

DETAILED DESCRIPTION:
We administered TAC(oxaliplatin,FUDR and MMC) 7 days before liver metastasis resection of colorectal cancer. The study endpoints were progression free survival and overall survival as evaluated by intent-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* age <= 75 years
* resectable liver metastasis
* remnant liver volume >= 70%
* without other organ metastasis or peritoneum metastasis
* without contradiction of cardiac and pulmonary diseases

Exclusion Criteria:

* age > 75 years
* unresectable liver metastasis
* remnant liver volume < 50%
* with other organ metastasis or peritoneum metastasis
* with contradiction of cardiac and pulmonary diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 5 years after operation

SECONDARY OUTCOMES:
overall survival | 5 years after operation

CONTACTS AND LOCATIONS:
Overall Officials: jianmin xu, MD, PHD, Principal Investigator — department of general surgery, zhongshan hospital, fudan university
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China